CLINICAL TRIAL: NCT03176992
Title: Surgicel® Versus Endometrial Ablation in the Management of Perimenpausal Heavy Menstrual Bleeding (HMB): Randomised Controlled Trial
Brief Title: Surgicel® & Endometrial Ablation in the Management of Perimenpausal Heavy Menstrual Bleeding
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moutaz Sherbini, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 250597
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Endometrial Hyperplasia
Keywords: ablation; surgicel
MeSH Terms: conditions — Endometrial Hyperplasia | interventions — Surgicel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Surgicel group (Active Comparator): 80 patients underwent formal curettage followed by insertion of 4 pieces of Surgicel inside the uterine cavity
  Interventions: Drug: SURGICEL®
- Thermal balloon ablation group (No Intervention): 80 patients underwent thermal balloon ablation using bipolar radiofrequency electrical energy (Novasure)
- Endometrial resection group (No Intervention): 80 patients underwent transcervical Hysteroscopic endometrial resection

INTERVENTIONS:
Drug: SURGICEL® — insertion of 4 pieces of Surgicel inside the uterine cavity after formal curettage
  Arms: Surgicel group

SUMMARY:
Two hundred & forty patients aged from 40 to 50 years - complaining of heavy menstrual bleeding that is unresponsive to hormonal lines of treatment & requesting conservative surgical approach- were randomized into 3 groups; group A (Surgicel group) in which 80 patients underwent formal curettage followed by insertion of 4 pieces of Surgicel inside the uterine cavity, group B (Thermal balloon ablation group) in which 80 patients underwent thermal balloon ablation using bipolar radiofrequency electrical energy (Novasure), group C (Endometrial resection group) in which 80 patients underwent transcervical Hysteroscopic endometrial resection.All patients were followed up over duration of 18 months following the procedure (at 3,6,12 & 18 months). Primary outcome included amenorrhea rates

DETAILED DESCRIPTION:
Two hundred & forty patients aged from 40 to 50 years complaining of heavy menstrual bleeding (i.e. pictorial blood loss assessment chart score >150) that is unresponsive to hormonal lines of treatment & requesting conservative surgical approach. Participants were randomized into 3 groups; group A (Surgicel group) in which 80 patients underwent formal curettage followed by insertion of 4 pieces of Surgicel inside the uterine cavity, group B (Thermal balloon ablation group) in which 80 patients underwent thermal balloon ablation using bipolar radiofrequency electrical energy (Novasure), group C (Endometrial resection group) in which 80 patients underwent transcervical Hysteroscopic endometrial resection. Randomization was done using computer generated random numbers.

Inclusion criteria included uterine length <12 cm, FSH level > 40 IU/L, normal Pap smear & benign endometrial pathology. Exclusion criteria included active form of PID, uterine scars, uterine malformation, uterine organic lesions (e.g., fibroids, polyps & Adenomyosis) & previous history of endometrial ablation. In addition, patients seeking fertility preservation, suffering coagulopathies or receiving anticoagulant treatments were excluded.

For all patients, full history was taken followed by complete physical examination (with emphasis on speculum examination to exclude cervical or vaginal wall lesions) & laboratory investigations (FSH, coagulation profile & routine preoperative investigations). History of Pap smear schedule was obtained and a Pap smear was scheduled if it was due. Transvaginal ultrasound (TVUS) was done using a 7.5 MHz vaginal probe of the General Electric Voluson E8 ultrasound unit (GE Healthcare Austria GmbH, Seoul, Korea) to assess uterine size and to exclude organic lesions of the uterus or ovaries. All participants were subjected to an endometrial biopsy (either before the procedure or intraoperatively followed by a frozen section). Patients, who were found to have atypical endometrial hyperplasia or endometrial malignancy, were excluded from the study.

In the Surgicel group (group A), each SURGICEL® (oxidized regenerated cellulose - Ethicon US, LLC.) knitted fabric (5 x 10 cm) was divided into four equal pieces. A formal cervical dilatation & curettage was done followed by packing the uterine cavity with the four SURGICEL® strips to ensure that the SURGICEL® is in contact with the basal endometrium all over the cavity.

In group B, Thermal balloon ablation was done using bipolar radiofrequency electrical energy (Novasure). The cervix was grasped with a tenaculum then dilated to 6 mm. The disposable device was inserted in the uterine cavity until the distal end of the sheath touches the fundus then withdrawn backwards approximately 0.5 cm. The cervical collar was slided forward until it forms a seal against the external cervical os. The ablation cycle starts automatically, upon successful completion of the cavity integrity assessment (CIA), & ends automatically as well. In group C, Transcervical hysteroscopic endometrial resection was done. Bipolar resectoscope is used & endometrium is resected in successive passes under direct hysteroscopic vision. Each pass of the U-shaped loop electrode removes a layer of tissue of approximately 3-5 mm.

All patients were followed up over duration of 18 months following the procedure (at 3,6,12 & 18 months). Primary outcome included amenorrhea rates & secondary outcomes included complication (intra- or post-operative), PBAC score (pictorial blood loss assessment chart score), dysmenorrhea rates, patient satisfaction & the need for re-intervention (hysterectomy).

ELIGIBILITY:
Inclusion Criteria:

* Heavy menstrual bleeding (i.e. pictorial blood loss assessment chart score >150) that unresponsive to hormonal lines of treatment & requesting conservative surgical approach.
* Uterine length <12 cm.
* FSH level > 40 IU/L
* Normal Pap smear
* Benign endometrial pathology

Exclusion Criteria:

* Active form of PID
* Uterine scars & uterine malformation.
* Uterine organic lesions (e.g., fibroids, polyps & Adenomyosis)
* Previous history of endometrial ablation.
* Patients seeking fertility preservation.
* Patients suffering coagulopathies or receiving anticoagulant treatments

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
amenorrhea rates | 18 months
  absence of menstruation

SECONDARY OUTCOMES:
PBAC score (pictorial blood loss assessment chart score) | 18 months
  chart consists of a series of diagrams representing lightly, moderately and heavily soiled towels and tampons.The participants complete the chart each menstrual period after clear instructions and explanation of how it should be used
dysmenorrhea rates | 18 months
  occurrence of painful menstruation
patient satisfaction | 18 months
  simple questions about decreasing duration & amount of menstrual blood & better quality of life
the need for re-intervention | 18 months
  hysterectomy

CONTACTS AND LOCATIONS:
Overall Officials: MOUTAZ ELSHERBINI, MD, Principal Investigator — Assistant professor of obstetrics and gynecology
Locations (1):
- kasr elaini hospital (Cairo university), Cairo, Egypt